CLINICAL TRIAL: NCT04111107
Title: Precision Medicine for Patients With Identified Actionable Mutations at Wake Forest Baptist Comprehensive Cancer Center (WFBCCC): A Pragmatic Trial-
Brief Title: Precision Medicine for Patients With Identified Actionable Mutations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left the institution and site decided not to continue the study
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00061185; WFBCCC 04519 (Other: IRB - Wake Forest University Health Science); P30CA012197 (NIH); NCI-2019-06802 (Other: Clinical Trials Reporting Program)
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Solid Tumor; Lymphoma; Multiple Myeloma; Malignant Neoplasm; Mutation Abnormality
MeSH Terms: conditions — Lymphoma; Multiple Myeloma; Neoplasms | interventions — Drugs, Investigational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Drug Administration Based on Next Gen Sequencing Report (Experimental): Investigators will select the first drug listed in the tumor analysis report for the first mutation listed in the tumor analysis report. However, If the subject has a medical contraindication to the first listed drug (according to the drug label) or the first listed drug cannot be obtained for the patient, the study team will select the next drug presented by the tumor sequencing report. Patients receive targeted therapy based on next generation sequencing report. Cycles repeat every 2, 4, or 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Investigational Agent; Other: Supportive Care Regimens; Diagnostic Test: Next Gen Sequencing Report

INTERVENTIONS:
Drug: Investigational Agent — Treatment will be administered on an inpatient or outpatient basis based on the type of medication selected. The investigatory will administer the drug as directed in the FDA approved label.
Other: Supportive Care Regimens — Supportive care regimens will vary depending on the type of drug that will be administered at the treating investigator's discretion.
Diagnostic Test: Next Gen Sequencing Report — 1) Next Gen Sequencing report obtained as Standard of Care within the past 12 months of enrollment date will be used. If more than one report exists in this time period, the most recent report will be used.

SUMMARY:
The goal of the current pragmatic trial is to evaluate the impact of a simple method of selecting a treatment approach for identified mutations on participants' progression free survival (PFS). The study also intends to collect information on barriers that investigators encounter when prescribing treatment options using the Next Generation Sequencing (NGS) reports. Additionally, patients' quality of life will be measured before, after, and during treatment.

Patients will be followed until death for monitoring survival study endpoints.

DETAILED DESCRIPTION:
Primary Objective:

• To estimate the progression-free ratio, as defined by the progression-free survival time on study treatment divided by the progression-free survival time on the last treatment received by patient, for an identified actionable mutation, who will be treated with an off-label treatment off label therapy based on a simplified selection methodology using the Next Generation Sequencing results.

Secondary Objectives:

* To estimate patient response rate on off-label treatments for actionable mutations based on Next Generation Sequencing results.
* To estimate overall survival (OS) for patients treated with off-label treatments for actionable mutations based on Next Generation Sequencing results.
* To describe the safety of using off-label or other experimental treatments for patients with actionable mutations based on Next Generation Sequencing results.

Exploratory Objectives:

* To describe health related quality of life in patients undergoing off-label treatment targeting genetic mutations, as measured by the PROMIS-29 Overall Health-Related Quality of Life, Including 4-Item Anxiety Subscale.
* Using the Satisfaction with Medical Decision Scale, to describe patient satisfaction with decision to pursue off-label treatment.
* To identify types of actionable mutations with available targeted treatment occurring in cancer patients.
* To characterize the historical treatment regimens for these patients relative to the targetable mutation.
* To describe patient clinical and demographic characteristics of those with actionable mutations based on Next Generation Sequencing results.
* To identify barriers to treatment based on Next Generation Sequencing results.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients at Wake Forest Baptist Comprehensive Cancer Center and its satellites who have next generation DNA sequencing results on their tumor biopsy or surgically resected tissue and/or blood samples and/or consent to the Wake Forest Comprehensive Cancer Center Precision Oncology Registry to use their information for research.
* Actionable mutation (defined as a mutation or gene amplification for which an off-label therapy is identified on the patient's NGS report for which NCCN guidelines do not recommend a specific treatment in the particular disease or for which there is no documentation in the patient's medical record of clinical data demonstrating lack of activity with the targeting of the specific mutation or amplification in the patient's specific disease) uncovered by the genomic sequencing of a tumor or those that have undergone liquid biopsy assay of their tumor genomic, performed by Wake Forest or another and who are medically able to receive targeted therapy based on those results.
* Sequencing on a sample collected within 3 months prior to registration is strongly encouraged but must have been performed within the 12 months prior to registration.
* Patients must have progressed through at least two lines of treatment, or are not candidates for or unwilling to receive any standard therapies. Patients who have received treatment on the present protocol who have progression of disease may be recruited to the trial for treatment using another targeted therapy provided that they fulfill the other criteria for participation in the trial. If a patient discontinues treatment on this protocol they can be considered for further participation in this trial provided they meet all of the eligibility criteria and are eligible for re-registration and re-consent.
* Eastern Cooperative Oncology Group (ECOG) of less than or equal to 3
* Life expectancy of greater than 6 weeks
* The effects of the drugs used for cancer treatment on the developing human fetus are unknown. For this reason and because of the possibility that the agents are teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* Patients who have had or will receive chemotherapy or radiotherapy to major bone marrow bearing sites within 2 weeks prior to receiving treatment on the study
* Patients who have not recovered from toxicity of prior treatment if such toxicity will preclude treatment with the proposed targeted agent.
* Patients may not be receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the targeted agent, breastfeeding should be discontinued if the mother is treated with the targeted agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2023-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Grant, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited between April 2020 and September 2022.
Period: Overall Study
Arm/Group | Drug Administration Based on Next Gen Sequencing Report
Started | 45
Completed | 34
Not Completed | 11
Not completed — Withdrawal by Subject | 6
Not completed — Declining Health | 5

BASELINE CHARACTERISTICS:
Arm/Group | Drug Administration Based on Next Gen Sequencing Report
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 36
  African American/Black | 8
  Hispanic/Latino | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45
Disease Site [Count of Participants; unit: Participants] — Not all participants had the same type of cancer. This measure is a grouping of the disease site. 'Head and Neck' includes hypopharynx, oropharynx, larynx, tonsil and tongue, salivary gland, thyroid, nasal cavity and brain. 'Other' includes ampulla of vater, intrahepatic bile duct, duodenum, prostate, rectum and skin.
  Participants
    Lung | 24
    Head and Neck | 13
    Other | 8

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Ratio
Description: Estimation of progression-free ratio defined as the duration of time from start of treatment to the time of progression divided by the duration of time from the last treatment received pre-trial to the time of progression on that treatment. The median progression-free ratio will be estimated with the range and a two-sided Wilcoxon Signed Rank test will be calculated to see if the progression free survival ratio is different from 1.0. This trial is powered to detect differences in the progression-free ratio for those with actionable mutations identified by NGS results and then treated with a targeted therapy. A hypothesized PFS ratio larger than 1.3 would suggest that the targeted therapy is doing better than the previous treatment received (not targeted), and we assume a null hypothesis PFS ratio of 1.0 (no difference).
Time Frame: From the start of treatment to the time of progression, death, or date of last contact, assessed up to 2 years
Population: For various reasons, 27 patients were not evaluable for the primary outcome. Five patients had no prior treatment but did have an actionable mutation to qualify them for inclusion in the study. Another ten patients were enrolled but never started treatment under this protocol. Nine patients started treatment but died prior to testing for best response and for progression. Two patients died with stable disease and one patient is alive with stable disease and no sign of progression .
Measure: Median (Full Range); unit: ratio
Arm/Group | Drug Administration Based on Next Gen Sequencing Report
Number analyzed (Participants) | 18
ratio | 0.73 [0.26 to 6.67]
Statistical Analysis 1: Comparison: Drug Administration Based on Next Gen Sequencing Report; H0: Progression-free ratio = 1; Test type: Other; p = 0.966, Wilcoxon signed rank (2 sided)

2. Secondary Outcome: Overall Survival
Description: Overall survival will be displayed using Kaplan-Meier curves with median survival times and 95% confidence intervals.
Time Frame: From the start of treatment to date of death or date of last contact, up to 2 years
Population: All enrolled participants, regardless of length of treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Drug Administration Based on Next Gen Sequencing Report
Number analyzed (Participants) | 45
months | 6.2 [4.3 to 8.8]

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events will be summarized in incidence tables by type for all patients who received at least one cycle of treatment.
Time Frame: Up to 30 days after treatment ends, up to 33 months
Population: Eleven patients did not begin treatment under this protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Administration Based on Next Gen Sequencing Report
Number analyzed (Participants) | 34
Participants | 34

4. Secondary Outcome: Response Rate
Description: Response rate will be estimated for all patients with corresponding 95% confidence intervals. Complete response is the disappearance of all target lesions and normalization of tumor marker level. Any pathological lymph nodes must have reduction in short axis to less than 10 mm. Partial response is at least 30% decrease in the sum of diameters of target lesions. Progressive disease is greater than 20% increase and a minimum 5 mm increase over the nadir. Stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Up to 30 days after treatment ends, up to 33 months
Population: Eleven patients did not receive study treatment (due to patient withdrawal or declining health) and ten patients died prior to evaluation for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Administration Based on Next Gen Sequencing Report
Number analyzed (Participants) | 24
Participants
  Partial Response | 1
  Stable Disease | 10
  Progressive Disease | 13
Statistical Analysis 1: Comparison: Drug Administration Based on Next Gen Sequencing Report; The proportion with a complete or partial response was estimated and an exact binomial confidence interval was calculated; Test type: Other — Single proportion was estimated; proportion = 4.2, 95% CI 2-sided [0.1 to 21.1] — exact binomial confidence interval

ADVERSE EVENTS:
Time Frame: Participants were followed for adverse events a minimum of 30 days after date of last study drug administration up to 33 months.
Arm/Group | Drug Administration Based on Next Gen Sequencing Report
All-Cause Mortality (participants affected / at risk) | 32/34
Serious Adverse Events (participants affected / at risk) | 18/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug Administration Based on Next Gen Sequencing Report (N=34)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Disease Progression (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
CPK increased (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Edema cerebral (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Recurrent laryngeal nerve palsy (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug Administration Based on Next Gen Sequencing Report (N=34)
Anemia (Blood and lymphatic system disorders) | 13 (34)
Heart Failure (Cardiac disorders) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 7 (9)
Vision decreased (Eye disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 6 (7)
Constipation (Gastrointestinal disorders) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 11 (12)
Dysphagia (Gastrointestinal disorders) | 3 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 12 (14)
Rectal- hemorrhage (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 13 (14)
Chills (General disorders) | 5 (5)
Edema limbs (General disorders) | 6 (7)
Fatigue (General disorders) | 19 (23)
Fever (General disorders) | 4 (6)
Malaise (General disorders) | 6 (6)
Pain (General disorders) | 4 (5)
Lung infection (Infections and infestations) | 3 (3)
Otitis media (Infections and infestations) | 2 (2)
Papulopustular rash (Infections and infestations) | 2 (2)
Pustular rash (Infections and infestations) | 2 (4)
Upper respiratory infection (Infections and infestations) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 6 (7)
Alanine aminotransferase increased (Investigations) | 7 (9)
Alkaline phosphatase increased (Investigations) | 15 (24)
Aspartate aminotransferase increased (Investigations) | 9 (12)
CPK increased (Investigations) | 3 (5)
Creatinine increased (Investigations) | 4 (6)
Lymphocyte count decreased (Investigations) | 22 (40)
Neutrophil count decreased (Investigations) | 8 (14)
Platelet count decreased (Investigations) | 14 (30)
Weight loss (Investigations) | 3 (3)
White blood cell decreased (Investigations) | 15 (28)
Anorexia (Metabolism and nutrition disorders) | 7 (8)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 14 (21)
Hypoalbuminemia (Metabolism and nutrition disorders) | 17 (28)
Hypocalcemia (Metabolism and nutrition disorders) | 15 (32)
Hypokalemia (Metabolism and nutrition disorders) | 5 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 10 (11)
Hyponatremia (Metabolism and nutrition disorders) | 19 (34)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 (7)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (7)
Cognitive disturbance (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 3 (4)
Dysgeusia (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 6 (10)
Lethargy (Nervous system disorders) | 4 (4)
Memory impairment (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Tremor (Nervous system disorders) | 2 (2)
Confusion (Psychiatric disorders) | 4 (4)
Urinary retention (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5)
Hypertension (Vascular disorders) | 8 (13)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/07/NCT04111107/Prot_SAP_001.pdf
  • Informed Consent Form (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT04111107/ICF_000.pdf